CLINICAL TRIAL: NCT04076514
Title: The Role of Central Neck Dissection in Stage N0 Papillary Thyroid Carcinoma
Acronym: pCND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Kamel Ali, resident, Assiut University
Other Study IDs: Ahmed1712
Record Dates: First submitted 2019-08-28; First posted 2019-09-03 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with node negative papillary thyroid carcinoma
  Interventions: Procedure: central neck dissection

INTERVENTIONS:
Procedure: central neck dissection — dissection of central cervical lymph node grope in low grade papillary thyroid cancer

SUMMARY:
The benefits of prophylactic central neck dissection (pCND) remain controversial in clinically node-negative (cN0) papillary thyroid carcinoma (PTC). This study main goal is to investigate benefits of prophylactic central neck dissection in clinically node-negative papillary thyroid carcinoma.

DETAILED DESCRIPTION:
Papillary thyroid carcinoma (PTC) is the most common type of differentiated thyroid carcinoma. Recurrence rate is still high. The standard management is total thyroidectomy. regional lymph node metastasis is noted in recurrent cases. Some studies stated benefits of central neck dissection in orevention of recurrence and others said there is no benefits. so prophylactic central neck dissection (pCND) remain controversial in clinically node-negative (cN0) papillary thyroid carcinoma (PTC).

ELIGIBILITY:
Inclusion Criteria:

* patients with papillary thyroid cancer with clinically node negative.

Exclusion Criteria:

* patients with clinical evidence of nodal metastases.
* patients with a previous history of thyroidectomy.
* patients with mixed-type papillary thyroid cancer.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with papillary thyroid carcinoma with clinically negative lymph node who undergo total thyroidectomy and central neck dissetion in assiut university hospital, department of general surgery.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
the incidence metastatic lymph node in patients with clinically node-negative thyroid carcinoma who underwent total thyroidectomy with central neck dissection | 12 months
  numbers of positive histopathological lymph node biopsies postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Kamel, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided